CLINICAL TRIAL: NCT06073600
Title: Randomized, Two-way, Two-period, Single Oral Dose, Open-label, Crossover, Bioequivalence Study to Compare Metformin / Vildagliptin Film Coated Tablets (1000 mg/50 mg) Versus Galvumet® Film Coated Tablets (1000 mg/50 mg)
Brief Title: Bioequivalence Study to Compare Metformin / Vildagliptin Versus Galvumet®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reseach Laboratory of Clinical and Experimental Pharmacology (Network)
Collaborators: La Société Arabe des Industries Pharmaceutiques-Tunisie (Unknown); Centre National Chalbi Belkahia de Pharmacovigilance-Tunisie (Unknown)
Responsible Party: Principal Investigator, Sameh Trabelsi, MD, Professor in Pharmacology, Reseach Laboratory of Clinical and Experimental Pharmacology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CNPVBE02-2022
Record Dates: First submitted 2022-06-21; First posted 2023-10-10 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Fed Conditions
Keywords: Bioequivalence; Metformin; Vildagliptin; Phase 1
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Intervention Model Description: This study is an open label, randomized, fed, single oral dose, two-treatment, two-sequence, and two-period crossover study with a washout interval of at least one week between dosing.
Who Masked: Outcomes Assessor
Masking Description: In this bioequivalence study, the bioanalysis, the pharmacokinetics and the statistical analysis will be blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First group of healthy volunteers (Experimental): The first group of healthy volunteers, defined by randomization
  Interventions: Drug: Metformin / Vildagliptin Reference Film Coated Tablets (1000 mg / 50 mg) (Galvumet®); Drug: Metformin / Vildagliptin Test Film Coated Tablets (1000 mg / 50 mg)
- Second group of healthy volunteers (Active Comparator): The second group of healthy volunteers, defined by randomization
  Interventions: Drug: Metformin / Vildagliptin Reference Film Coated Tablets (1000 mg / 50 mg) (Galvumet®); Drug: Metformin / Vildagliptin Test Film Coated Tablets (1000 mg / 50 mg)

INTERVENTIONS:
Drug: Metformin / Vildagliptin Reference Film Coated Tablets (1000 mg / 50 mg) (Galvumet®) — The subjects randomly received a single oral administration of Metformin / Vildagliptin Film Coated Tablets (1000 mg / 50 mg).
  Other Names: Galvumet®
Drug: Metformin / Vildagliptin Test Film Coated Tablets (1000 mg / 50 mg) — The subjects randomly received a single oral administration of Metformin / Vildagliptin Film Coated Tablets (1000 mg / 50 mg).
  Other Names: BiGalvine

SUMMARY:
The aim of this study is to assess bioequivalence between a single oral dose from the test product Metformin / Vildagliptin tablets (1000 mg as metformin hydrochloride / 50 mg as vildagliptin) manufactured by Pharmaceutical Arab Industries Society, Tunisia versus the reference product Galvumet® tablets (1000 mg as metformin hydrochloride / 50 mg as vildagliptin) manufactured by Novartis.

This study also aims to monitor the safety of the subjects. This study is an open label, randomized, fed, single oral dose, two-treatment, two-sequence, and two-period crossover study with a washout interval of at least one week between dosing.

Eighteen (18) Tunisian subjects will be enrolled for this study. Subjects will be healthy volunteers, adults, aged between eighteen to fifty (18-50) years, (both inclusive), within the accepted limits for body height & weight and meeting the selection criteria for this study.

DETAILED DESCRIPTION:
The aim of this study is to assess bioequivalence between a single oral dose from the test product Metformin / Vildagliptin tablets (1000 mg as metformin hydrochloride / 50 mg as vildagliptin) manufactured by Pharmaceutical Arab Industries Society, Tunisia versus the reference product Galvumet® tablets (1000 mg as metformin hydrochloride / 50 mg as vildagliptin) manufactured by Novartis.

This study also aims to monitor the safety of the subjects. This study is an open label, randomized, fed, single oral dose, two-treatment, two-sequence, and two-period crossover study with a washout interval of at least one week between dosing.

Eighteen (18) Tunisian subjects will be enrolled for this study. Subjects will be healthy volunteers, adults, aged between eighteen to fifty (18-50) years, (both inclusive), within the accepted limits for body height & weight and meeting the selection criteria for this study.

Products under investigation for this study:

Test Product: Metformin / Vildagliptin tablets (1000 mg as metformin hydrochloride / 50 mg as vildagliptin) manufactured by Pharmaceutical Arab Industries Society, Tunisia.

Reference Product: Galvumet® tablets (1000 mg as metformin hydrochloride / 50 mg as vildagliptin) manufactured by Novartis.

Metformin and vildagliptin are two oral antidiabetic drugs. Metformin belongs to biguanide class. Vildagliptin is a selective inhibitor of dipeptidyl peptidase-4 (DPP-4).

Metformin and vildagliptin are indicated as an adjunct to diet and exercise to improve glycemic control in adults with type two diabetes mellitus.

This study will be conducted according to the principles of Good Clinical Practice (GCP) that have their origins in the Declaration of Helsinki.

This study will be subject to the review and approval of Persons Protection Committee and of Pharmacy and Medicine Department.

Subjects will not be recruited without obtaining their informed consent. Subjects will be covered for adverse events through an insurance company. Subjects will be housed in each study period at least 12 hours before dose administration and until 36 hours after dosing.

Subjects will be in a sitting position on chairs for the first 4 hours that follow the dose.

After an overnight fast of ten to twelve (10-12) hours and in the morning of the second day of each study period (day 2), a standard high-fat breakfast (800-1000 calories) will be served to subjects, thirteen (30) minutes before dosing.

At 08:00 am, the study products will be administered orally in a randomized fashion with 240 ± 2 mL warm 20% glucose solution.

During each period of the study, 21 blood samples of 7 mL each will be collected (via an indwelling cannula into lithium heparin tubes) according to the following schedule: Pre dosing (zero time) and 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 2.5, 3.00, 3.50, 4.00, 4.5, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 14.00, 24.00 & 36.00 hours post dosing.

After collection, the blood samples will be placed in an ice bath or other chilling device until centrifugation.

Before each period of the study, 21 mL blood sample will be collected for bio-analytical purposes.

A blood sample of 3 mL may be needed for a possible control. Samples will be centrifuged at 4000 round per minute for 5 minutes at 10°C. Supernatant plasma will be transferred to pre-labeled polypropylene Eppendorf tubes and stored in freezers at nominal temperature of -20 C unless otherwise advised by the stability studies on samples.

Samples from all subjects will be analyzed at the bio-analytical site of the National Center of Pharmacovigilance according to validated in-house procedure using validated Liquid Chromatography-Mass Spectrometry Tandem method for the plasma concentrations of metformin & vildagliptin.

Primary end points would be obtaining the following pharmacokinetic parameters for metformin & vildagliptin: Cmax, Air Under Cover (AUC) 0 - t & AUC 0 - ∞.

Secondary end points would be obtaining the following pharmacokinetic parameters for metformin & vildagliptin: Tmax, T half & K elimination (λz).

Statistical analysis of primary endpoints will include descriptive statistics, Analysis of Variance (ANOVA), and Confidence Interval (CI). The average bioequivalence of the products is concluded if the two-sided 90 % CI for the test to reference ratio of the population means is within 80.00 - 125.00 % for each of the Ln-transformed data of the following primary end points for metformin & vildagliptin: Cmax, AUC 0 - t & AUC 0 - ∞ and if there were no safety concerns and both products were well tolerated by the study subjects.

ELIGIBILITY:
Inclusion Criteria:

A. The subject is aged between eighteen to fifty years (18 - 50), both inclusive.

B. The subject is within the limits for his height & weight as defined by the body mass index (BMI) range (18.5 - 30.0 Kg/m2).

C. The subject is able to understand and willing to sign the Informed Consent Form.

D. The subject has completed his Coronavirus 19 vaccination schedule. E. The subject is willing to undergo the necessary medical examinations pre- during & post-study.

F. There is no evidence of psychiatric disorder, antagonistic personality, and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.

G. The results of medical history, physical examination, vital signs, conducted medical laboratory tests & ECG recording are normal as determined by the investigator.

H. The subject tested negative for Hepatitis B (HBsAg) and Hepatitis C (HCVAb). I. For female subjects: negative pregnancy test and the woman is using two reliable contraception methods and should be non-lactating.

Non-inclusion Criteria:

A. The subject is a heavy smoker (more than 10 cigarettes per day). B. The subject has a history of or concurrent abuse of alcohol. C. The subject has a history of or concurrent abuse of illicit drugs. D. The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds.

E. The subject is vegetarian. F. The subject has suffered an acute illness within seven (7) days before first dosing (declared before inclusion).

G. The subject has been hospitalized within three (3) months before the study. H. The subject has taken a prescription medication within two weeks or even an over-the-counter product (OTC) within seven (7) days before first dosing.

I. The subject has taken grapefruit containing beverages or foodstuffs within seven (7) days before first dosing (declared before inclusion).

J. The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.

K. The subject has been participating in any clinical study (e.g. PKs, BA and BE studies) within the last 80 days prior to the present study.

L. The subject has donated blood within 80 days before first dosing.

Exclusion Criteria:

A. The subject has suffered an acute illness within seven (7) days before dosing (declared after inclusion).

B. The subject has been hospitalized during the study. C. The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two (2) days before dosing and until 12 Hrs after dosing in both study periods.

D. The subject has taken a prescription medication within two (2) weeks or even an OTC within seven (7) days before first dosing and any time during the study unless otherwise judged acceptable by the investigator.

E. The subject has taken grapefruit containing beverages or foodstuffs within seven (7) days before dosing (declared after inclusion) and any time during the study.

F. The subject underwent a radiological examination with an injection of Iodinated Contrast Media within 48 hours before first dosing.

G. The subject has a positive Covid-19 rapid test.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-11-13 (Actual)

PRIMARY OUTCOMES:
Cmax | 2 - 4 Hours
  obtaining the following pharmacokinetic parameters for metformin & vildagliptin: Cmax.
AUC 0 - t | 0 - 24 Hours
  obtaining the following pharmacokinetic parameters for metformin & vildagliptin: AUC 0 - t.

SECONDARY OUTCOMES:
Tmax | 2 - 4 Hours
  obtaining the following pharmacokinetic parameters for metformin & vildagliptin: Tmax
T half | 7 days
  obtaining the following pharmacokinetic parameters for metformin & vildagliptin: T half
K elimination (λz) | 7 days
  obtaining the following pharmacokinetic parameters for metformin & vildagliptin: K elimination (λz)

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Trabelsi, Principal Investigator — Research Laboratory of Clinical and experimental Pharmacology LR16SP02
Locations (1):
- Centre National Chalbi Belkahia de Pharmacovogilance, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No